CLINICAL TRIAL: NCT04610918
Title: Comparing Body Composition Assessment Methods, Evaluating Physical Activity and Strength in Children With Intestinal Failure: Building a Framework for More Personalized and Holistic Care in Pediatric Intestinal Failure
Brief Title: Comparing Body Composition Assessment Methods
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Rare Disease Foundation (Unknown)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Principal Investigator, The Hospital for Sick Children
Other Study IDs: 1000069821
Record Dates: First submitted 2020-10-06; First posted 2020-11-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Body Composition; Gastrointestinal Failure; Pediatric ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases - Pediatric Intestinal Failure Patients: DXA BIA Skin fold measurements Strength tests Physical activity monitoring
- Controls: BIA Skin fold measurements Strength tests Physical activity monitoring

SUMMARY:
Background: Improvement in clinical care has resulted in longer life expectancy of children with intestinal failure (IF). However, recent data indicate that their body composition (BC) is abnormal with a relatively high fat mass (FM) and low fat free mass (FFM). Abnormal BC is linked to poor prognosis and increased length of hospital stay; yet BC is not assessed in pediatric clinical practice. Instead, growth charts which lack sensitivity to detect changes in BC are used. Physical activity (PA) is the most important predictor of FFM and increased PA contributes to decreased FM. Decreased PA in childhood is associated with increased FM and decreased FFM which are linked to diabetes and cardiovascular disease in adulthood. Dual-energy X-ray Absorptiometry (DXA) is considered the reference method for measuring BC in the clinical setting but it is expensive and not suitable for routine use. Bioelectrical Impedance Analysis (BIA) on the other hand is relatively inexpensive and non-invasive but needs to be validated for use in patients with IF. Objectives: 1) validate BIA against DXA as a clinical tool for monitoring changes in BC in children with IF, 2) quantify PA levels using activity counts from accelerometers and 3) assess strength. Design: 1-18 years, with IF followed by the intestinal rehabilitation program at SickKids. All subjects receiving a DXA for routine clinical monitoring are eligible. BIA and muscle strength will be measured in clinic. Demographic data and IF related factors including height, weight, PN prescription, age, diagnosis, bowel length and length of time off PN for those who have achieved enteral autonomy will be obtained. DXA measurement will be done by Diagnostic Imaging at SickKids. Patients will be fitted with an accelerometer to be worn for 7 days. Statistics: Differences between sexes will be assessed by t test. Relationship between PA and BC, and BC and muscular strength will be assessed by linear regression analysis. Agreement between DXA and BIA will be assessed using a Bland-Altman test. Significance will be set at p<0.05. Significance: This study has the potential to establish BIA as a convenient clinical tool to assess BC and provide a more accurate basis for nutritional and PA prescriptions to optimize long-term outcomes and quality of life in IF patients.

DETAILED DESCRIPTION:
METHODOLOGY:

Subjects:

Participants with IF will be recruited from patients followed by our multidisciplinary intestinal rehabilitation program at SickKids.

Exclusion criteria: patients who are wheelchair bound or non-weight bearing, those unwilling to participate.

Methods:

An annual DXA is ordered for all our patients beginning at 1-year of age as part of routine clinical monitoring. On the day of the scheduled DXA, FFM using BIA, FM using Skinfolds and muscle strength will be measured in clinic. After DXA measurement, patients will be fitted with an accelerometer to be worn for 7 days.

Body composition: 3 methods - BIA, Skinfolds & DXA

Whole body and segmental BIA (leg, trunk and arm) will be taken on the right side of the body using a fixed frequency analyzer (50kHz) (BIA model 101A: RJL Systems). Resistance (R) and reactance (Xc) measurements will be made using 4-terminal bioelectrical impedance analyzer according to the manufacturer's recommendations after 10 hour overnight fasting for patients on enteral nutrition. Three readings R and Xc (in) will be taken from each subject. Patients on parenteral nutrition (PN) will be prescribed a standard fluid intake of 130 mls/kg and be cycled off PN for 3 hrs before measurement of BC. Body composition will also be assessed by BIA in clinic and DXA (GE-Lunar DPS Pro (EG Healthcare, Waukesha, WI, USA), at the Radiology Department, SickKids as part of routine annual clinical monitoring.

Four SF thicknesses (triceps, biceps, subscapular, and super iliac) will measured to the nearest 1mm with a Harpenden caliper to obtain estimates of fat mass.

Anthropometric & IF related factors: Data will be collected on PN prescription, % of calories on PN and enteral nutrition, number of months weaned of PN (if off PN), age, sex, diagnosis, weight and height.

Physical activity level:

Physical activity will be measured by accelerometry using the Actigraph GT3X accelerometer for measuring activity counts. It provides quantitative information regarding vertical acceleration of the trunk, and lower body parts at specified time intervals and can be used to evaluate frequency, intensity and duration of PA. Their small size and robust design make them an excellent alternative for use in children. They are less burdensome relative to heart rate monitors and capable of detecting the intermittent activity patterns characteristic of children.

Participants will be asked to wear the accelerometer for 7 consecutive days, including two weekend days during waking hours except when participating in water related activities (e.g., showering, swimming). The accelerometer will be worn on an elastic belt on the right hip, above the iliac crest. Each subject will receive a call by a research coordinator to remind them to wear the monitor. Subjects will also be given a handout that will include common solutions to potential barriers for wearing the monitor along with a prepaid envelope to return the accelerometer at the completion of the 7 days. Data from the accelerometers will be downloaded and analyzed with the manufacturer's software.

Muscle strength

In this study, objective measures will be used to assess both functional strength and specific muscle strength of the participants. The Bruininks-Oseretsky Test of Motor Proficiency-2 (BOT-2) is norm referenced and designed to measure gross and fine motor skills in children and youth 4-21 years of age. It is a widely accepted test with a reliable and efficient measure of motor proficiency. The strength subtest will be utilized in this study and is designed to measure functional strength. Children will be tested on their grip strength using a Jamar 5030J1 dynamometer. Specific muscle strength of select arm and leg muscles will also be measured clinically by a physiotherapist.

Subjects:

Patient with intestinal failure:

Patients with IF will undergo all tests as described above. Before clinic visit, patients will be contacted by the person preparing for clinic (a study team member) and the study will be introduced to the parents or child by a member of the health care team. If parents are interested, the study will be further explained in clinic and any questions answered by a study team member. The same person will obtain informed consent/assent (study team member but not a member of the health care team) Patients will be recruited in clinic.

All patients with IF followed by the GIFT team at the hospital and aged 1-18 years will be eligible to participate except those who are wheel chair bound.

Control participants:

Healthy control participants will be recruited by posting flyers in common areas at the Hospital for Sick Children and the PGCRL. Contact information for the study team member accepting enquire will be included on the flyer. These postings will be negotiated through Public Affairs. Healthy controls will also be recruited through families of patients with IF and children of staff members and other colleagues at the Hospital for Sick Children. Two healthy controls will be recruited for each case.

Healthy controls will be age, race and sex matched. Age will be matched within ±2 months for subjects between 1-3 years and within ±6 month for those 4 years and above.

Both IF patents and controls will be fitted with an accelerometer and sent home to wear it for 7 days. A stamped and addressed envelope will be given to mail the accelerometer back to the hospital for those patient who live outside of the GTA. For those residing within the GTA, the accelerometers will be picked up from their homes or an arranged location by study team members.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Intestinal Failure will be recruited from patients followed by our multidisciplinary intestinal rehabilitation program at SickKids. A total of about 133 patients are seen annually.
* Healthy controls will be age, race and sex matched. Age will be matched within ±2 months for subjects between 1-3 years and within ±6 month for those 4 years and above.
* Aged 1-18 years

Exclusion Criteria:

* patients who are wheelchair bound or non-weight bearing, those unwilling to participate.

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients with Intestinal failure (IF) which is the inability of the gastrointestinal tract to absorb adequate fluid and nutrients for growth and maintenance due to disease associated loss of absorption.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Body composition of children with intestinal failure compared with healthy controls. | 11/1 2020 - 10/1/2023
  measurement of fat and fat-free mass by BIA and DXA

SECONDARY OUTCOMES:
To measure physical activity and strength of children with intestinal failure compared with healthy controls. | 11/1 2020 - 10/1/2023
  Strength will be measured in children with intestinal failure and healthy age and sex matched controls using standard instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Courtney-Martin, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yanchis D, So S, Patterson C, Belza C, Garofalo E, Wong-Sterling S, Silva C, Avitzur Y, Wales PW, Hulst JM, Kong D, Xu L, Li Y, Courtney-Martin G. Reduced strength is associated with abnormal body composition in children with a history of intestinal failure. J Pediatr Gastroenterol Nutr. 2026 Feb;82(2):615-624. doi: 10.1002/jpn3.70307. Epub 2025 Dec 9. PMID 41363022